CLINICAL TRIAL: NCT02196298
Title: A Randomized Cross-over Clinical Trial Comparing the Impact of the Lokomat® Gait Training System With a Gait-related Physiotherapy Program in Children With Cerebral Palsy
Brief Title: A Randomized Trial Comparing the Lokomat® With a Gait-related Physiotherapy Program in Children With Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: CIBC Children's Foundation (Unknown)
Responsible Party: Principal Investigator, Virginia Wright, Senior Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-293
Record Dates: First submitted 2014-04-09; First posted 2014-07-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cerebral Palsy
Keywords: physical therapy; gait; pediatric rehabilitation; gross motor function; participation
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lokomat (Experimental): 16 sessions in total, 30 minutes each plus set-up time followed by 5 minutes of overground walking. Provided by study PT twice weekly for a period of 8 weeks to maximum of 10 weeks.
  Interventions: Device: Lokomat
- Physiotherapy (Active Comparator): 16 sessions, 35 minutes. Provided by study PT twice weekly for a period of 8 weeks to maximum of 10 weeks.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: Lokomat — 16 sessions in total, 30 minutes each plus set-up time followed by 5 minutes of overground walking. Provided by study PT twice weekly for a period of 8 weeks to maximum of 10 weeks.
  Other Names: Lokomat®Pro Pediatric Orthoses
  Arms: Lokomat
Other: Physiotherapy — 16 sessions, 35 minutes. Provided by study PT twice weekly for a period of 8 weeks to maximum of 10 weeks.
  Arms: Physiotherapy

SUMMARY:
The Lokomat is a robotic treadmill gait trainer that is used to help people who have neurologic conditions walk better. Early research with children with cerebral palsy (CP) shows that it may help to improve walking skills. The purpose of this two-group randomized study is to compare Lokomat training to regular physiotherapy (PT) as far as impact on walking abilities and related function. The primary (alternate) hypothesis is that children will improve more with Lokomat training in terms of gross motor skills and walking endurance.

The investigators are enrolling 40 ambulatory children who are ages 5 to 12 years, have CP and are in Gross Motor Function Classification System (GMFCS) Level II (n=20) or III (n=20). In this crossover randomized clinical trial (RCT), whether PT or Lokomat intervention is done first is decided by an independent randomization process that occurs after the first baseline assessment. In the Lokomat phase, children receive 8 to 10 weeks of twice weekly therapy for a maximum of 16 sessions. Each session is 35 minutes plus the time needed for set-up. The 35 minute PT program is also given twice weekly for 8 to 10 weeks for a maximum of 16 sessions, and focuses on a menu-based strength, co-ordination, fitness, walking and balance activities. There is a 6 week break between the Lokomat and PT interventions.

Each child has four study assessments during their ~6 months in the study. The first assessment is done before starting the Lokomat or physiotherapy phase. The second happens after the first intervention has finished. The child then has a 6-week break period. The third assessment is done at the end of this break, and the fourth occurs after the second intervention. The PT assessor who does these assessments will not be the same as the PT who gives the intervention. The assessor is blinded to the child's intervention phase and previous assessment results. The primary outcome measures are the Gross Motor Function Measure and 6 minute walk test. Secondary measures evaluate gait, functional abilities, participation, health related quality of life and individualized goals.

The randomized aspect of the study lets us look at outcome differences between children for Lokomat and PT within their first intervention phase (n=20/group). The cross-over phase evaluates within-child outcomes across the two phases. A qualitative component is concurrently underway to examine child/parent experiences and their views of Lokomat outcomes.

DETAILED DESCRIPTION:
No further information

ELIGIBILITY:
Inclusion Criteria:

* age 5 to12 years inclusive
* assessed as GMFCS Levels II or III
* able to follow testing instructions, and participate in a minimum of 30 minutes of active PT
* able to reliably signal pain, fear and discomfort
* have passive range of motion (ROM) of hips and knees within minimum range requirement for Lokomat (hip and knee flexion contracture < 10 degrees, and knee valgus < 40 degrees)
* client of Child Development Program at Holland Bloorview
* able to commit to attendance of twice weekly for eight weeks (to support the primary efficacy analysis).

Exclusion Criteria:

* a fixed knee contracture > 10 degrees, knee valgus >40 degrees such that robotic leg orthosis will not be adaptable to lower limbs
* hip instability/subluxation > 45%
* orthopaedic surgery within the last 9 months (muscle) or 12 months (bone)
* Botulinum toxin-A (BTX-A) injections to lower limb in the last 4 months
* inability to discontinue BTX-A for period of 6 months (during trial) due to concerns about ROM or pain
* severe spasticity may be a contraindication
* any weightbearing restrictions
* seizure disorder that is not controlled by medication (if on medication, must not have had a seizure in the last 12 months)
* open skin lesions or vascular disorder of lower extremities
* not able to co-operate or be positioned adequately within the Lokomat as shown during the two Lokomat fitting/acclimatisation sessions
* not prepared or unable to discontinue a regular therapy intervention during the course of the trial
* involved in another intervention study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in motor function on Gross Motor Function Measure (GMFM-66) at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Stand and Walk items of the GMFM-66. Gold standard measure of foundational gross motor skills in children with CP.

SECONDARY OUTCOMES:
Change from baseline in walk speed on the Six-minute walk test at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Used as the co-primary outcome measure. Standardized 6 minute walk test (with shoes, orthoses, walking devices as required) to determine distance covered (capability measure). Well-validated in pediatric CP.
Change from baseline in advanced motor skills on the Challenge Module at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Just for children in GMFCS Level II. This is a new published measure of advanced motor skills.
Change from baseline in activity and participation on the Activities Scale for Kids at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Well-validated measure of physical functional ability in children. Child (if 8+ years) or parent-report questionnaire
Change from baseline in quality of life on the KidScreen Questionnaire at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Measure of health-related quality of life. Questionnaire completed by children 8+ years or parents of younger children.
Change from baseline in participation on the Children's Assessment of Participation and Enjoyment (CAPE) at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Using the physical activity and sport sections of this parent-report questionnaire to gain picture of areas/extent of participation in these areas.
Change from baseline in gait kinematics as measured on the GaitRite evaluation system at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Time distance parameters of gait via GaitRite system
Change from baseline in Gait quality as measured on an observational gait scale at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Gait pattern as evaluated via observational gait scale, rating from video of child's walking
Change from baseline in targeted goal abilities as measured by Goal Attainment Scaling (GAS) at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Three to five individualized walking-based activity/participation goals set with child/parent/treating PT at baseline 1 and reset at baseline 2. Evaluated by treating PT with child/parent input at post-intervention 1 and 2
Change from baseline in targeted goal abilities and satisfaction with performance as measured by the Canadian Occupational Performance Measure at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Three to five individualized walking-based activity/participation set at baseline 1 and 2 with assessor and child/parent, and re-evaluated by child/parent at post-intervention assessment 1 and 2. Used by treating PT to formulate GAS goals
Change from baseline in movement quality as measured by the Quality Function Measure (QFM) at week 8 | Baseline, 8 weeks (repeated in same manner after crossover)
  Companion measure to the GMFM-66 to assess alignment, co-ordination, dissociated movement, stability and weight shift. Rated by PT assessor from GMFM video. Recently validated.

OTHER OUTCOMES:
Assessment of mastery motivation using the Dimensions of Mastery Questionnaire at the first baseline | Baseline 1 only
  This measure of a child's motivation and persistence with difficult tasks is a measure of traits rather than outcome. Not expected to change so being used instead as a possible predictor of outcomes. Questionnaire completed by child (if 8+ years) or parent-report questionnaire
Monitoring of range of motion (ROM) of hip, knee and ankle | baseline, 4 weeks, 8 weeks (repeated in same manner after crossover)
  Hip, knee, ankle - passive ROM
Body pain | participants will be followed at each treatment session for the duration of the study, an expected average of 16 weeks (8 weeks in the Lokomat arm and 8 weeks in the PT arm)
  Use of FACES pain scale and body diagrams to show areas of pain (skin and musculoskeletal and other)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Wright, PT, PhD, Principal Investigator — Holland Bloorview Kids Rehabiltation Hospital; Darcy Fehlings, MD, MSc, Principal Investigator — Holland Bloorview Kids Rehabiltation Hospital
Locations (1):
- Holland Bloorview Kids Rehabiltation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hilderley AJ, Fehlings D, Lee GW, Wright FV. Comparison of a robotic-assisted gait training program with a program of functional gait training for children with cerebral palsy: design and methods of a two group randomized controlled cross-over trial. Springerplus. 2016 Oct 28;5(1):1886. doi: 10.1186/s40064-016-3535-0. eCollection 2016. PMID 27843743
- [Background] Phelan SK, Gibson BE, Wright FV. What is it like to walk with the help of a robot? Children's perspectives on robotic gait training technology. Disabil Rehabil. 2015;37(24):2272-81. doi: 10.3109/09638288.2015.1019648. Epub 2015 Apr 9. PMID 25856202
- [Background] Beveridge B, Feltracco D, Struyf J, Strauss E, Dang S, Phelan S, Wright FV, Gibson BE. "You gotta try it all": Parents' Experiences with Robotic Gait Training for their Children with Cerebral Palsy. Phys Occup Ther Pediatr. 2015;35(4):327-41. doi: 10.3109/01942638.2014.990547. Epub 2014 Dec 20. PMID 25529412
- See also: Website of facility where trial is occurring. Investigators' lab sites are also on that website — http://www.hollandbloorview.ca